CLINICAL TRIAL: NCT02242591
Title: Effect of Adductor Canal Block vs. Placebo on Muscle Strength, Mobilisation and Pain on the First Post-operative Day After Total Knee Arthroplasty
Brief Title: Effect of Adductor Canal Block vs. Placebo on Muscle Strength, Mobilisation and Pain After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ulrik Grevstad (Other)
Responsible Party: Sponsor-Investigator, Ulrik Grevstad, Consultant, MD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-002245-21
Record Dates: First submitted 2014-09-12; First posted 2014-09-17 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Knee Replacement Arthroplasty
Keywords: Knee surgery; Saphenous nerve; Perineural block; Adductor Canal Block; Postoperative Pain; Mobilization
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride; Sodium; Chlorides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACB_active/placebo (Active Comparator): Patients will receive the first ACB with a active drug, 30 ml bolus Ropivacaine 7,5 mg/ml at T0. First outcome measurement are made one hour after the first ACB, prior to their second ACB. At T60 (60 minutes after T0), patients will receive their second ACB with the placebo drug, 30 ml bolus Saline and outcome measures performed again at T120(120 minutes after T0).
  The measurements for baseline and outcome will be made in following order:
  VAS pain score at rest - VAS pain score during active flexion of the knee - Muscle strength - TUG test - Highest VAS pain score during TUG test
  Interventions: Drug: Ropivacaine 7,5 mg/ml; Drug: Saline
- ACB_placebo/active (Placebo Comparator): Patients will receive the first ACB with placebo, 30 ml isotonic saline at T0. First outcome measurement are made one hour after the first ACB, prior to their second ACB. At T60(60 minutes after T0), patients will receive their second ACB with the ropivacaine 7,5 mg/ml 30 ml and outcome measures performed again at T120(120 minutes after T0).
  The measurements for baseline and outcome will be made in following order:
  VAS pain score at rest - VAS pain score during active flexion of the knee - Muscle strength - TUG test - Highest VAS pain score during TUG test
  Interventions: Drug: Ropivacaine 7,5 mg/ml; Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine 7,5 mg/ml
  Other Names: Product name: Ropivacain "Fresenius Kabi"; Ropivacainhydrochloridmonohydrat; Importet to Denmark by Fresenius Kabi AB; Injection mixture
Drug: Saline
  Other Names: Product name: Natriumklorid "Fresenius Kabi" 9 mg/ml; Sodium 9g/l; Electrolyte content: Na+ 154 mmol/l; Cl- 154 mmol/l; Infusion mixture

SUMMARY:
The purpose of this study is to evaluate the effect of adductor canal block (ACB) vs. placebo on muscle strength, mobility and pain on the first postoperative day after total knee alloplastic (TKA).

DETAILED DESCRIPTION:
Patients will be included on the first day after TKA surgery and randomized in two groups. Each group will receive 2 ACB with a 1 hour interval, one ACB with an active drug, Ropivacaine, and another ACB with a placebo drug, Saline.

At T0, arm ACB_active/placebo will receive the active ACB with Ropivacaine followed by the placebo ACB at T60 (60 minutes after T0).

At T0, arm ACB_placebo/active will receive the placebo ACB with Saline followed by the active ACB with Ropivacaine at T60 (60 minutes after T0).

Outcome measurements will be made at T60, 1 hour after the first ACB, and the difference in outcome between the groups will be compared.

Baseline values will be measured prior to the first ACB. Final measurements at T120 (120 minutes after the initial ACB), will determine if the differences between the groups are eliminated, since both groups then have received an active ACB.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a Total Knee Arthroplasty surgery within 2 days (1.postoperative day on inclusion)
* Written informed consent.
* ASA 1-3

Exclusion Criteria:

* Non-cooperative patients
* Patients who have already had a peripheral or central block post surgery.
* Patients who are not able to perform a TUG test pre surgery.
* Patients who do not understand or speak Danish.
* Patient who are allergic to the drugs used in this research.
* Patients with alcohol- or drug abuse - determined by investigator.
* Patients with peripheral sensory neuropathy in their lower extremities.
* Pregnant patients.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Difference between groups in muscle strength of the quadriceps femoris muscle. | 60 minutes after first ACB (T60)
  Muscle strength is assessed as maximum voluntary isometric contraction (MVIC) using a hand-held dynamometer.3 consecutive measurements will be made and the average used. Results for each group will be presented as percentage of baseline values. The primary outcome is the difference in MVIC between the groups.

SECONDARY OUTCOMES:
Difference between groups in muscle strength of the quadriceps femoris muscle. | 120 minutes after initial ACB (T120)
  Same as primary outcome
VAS pain scores at rest | 60 minutes after the initial ACB (T60) and 120 minutes after initial ACB (T120)
  Pain at rest (VAS 0-100 mm) one hour after the first and second ACB. Results will be compared between the two groups.
  VAS pain scores at rest will be inquired before any other outcome measurements.
VAS pain score during TUG test. | 60 minutes after the initial ACB (T60) and 120 minutes after initial ACB (T120
  Highest VAS (0-100 mm) pain score during TUG test will be inquired for each TUG test. Results will be compared between the two groups.
Timed Up and Go(TUG) test | 60 minutes after the initial ACB (T60) and 120 minutes after initial ACB (T120
  Time (seconds) to complete a TUG test measured one hour after the first and second ACB. Results will be compared between the two groups.
VAS pain scores during 45 degrees active flexion of the knee | 60 minutes after the initial ACB (T60) and 120 minutes after initial ACB (T120
  Specification of pain (VAS 0-100 mm) during 45 degrees active flexion of the knee one hour after first and second ACB. Results will be compared between the two groups.
Sub-group analysis of muscle strength and mobility acconding to baseline VAS during active flexion of the knee prior to the first block | 60 minutes after first ACB (T60)
  According to their specified VAS (0-100 mm) pain score during active flexion of the knee prior to the first block, patients will be divided into two groups. Group 1 VAS 0-59 mm and group 2 with VAS 60-100 mm. Results within the two groups will be compared: e.g is there a difference in MVIC in the subgroup of patients scoring VAS 0-59 during active knee flexion at baseline? and is this difference larger in the subgroup of patients scoring VAS 60-100?

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Grevstad, MD, Principal Investigator — Gentofte Hospital
Locations (1):
- Gentofte Hospital, Hellerup, Denmark